CLINICAL TRIAL: NCT06642545
Title: A Randomized, Open-label, Controlled, Multicenter Phase II Study to Evaluate the Efficacy and Safety of Disitamab Vedotin Combined With RC148 Versus Albumin-bound Paclitaxone Alone or in Combination With Toripalimab in Subjects With HR-negative, HER2-low Expressing Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: Efficacy and Safety Study of Disitamab Vedotin + RC148 vs. Albumin-Paclitaxone ± Toripalimab in HR-/HER2-low Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C036
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin +RC148 (Experimental)
  Interventions: Drug: Disitamab Vedotin; Drug: RC148
- Albumin-bound Paclitaxone OR Albumin-bound Paclitaxone +Toripalimab (Active Comparator)
  Interventions: Drug: Albumin-bound Paclitaxone; Drug: Toripalimab

INTERVENTIONS:
Drug: Disitamab Vedotin — Disitamab Vedotin 2.0mg/kg,intravenous infusion, every 2 weeks
  Other Names: RC48
  Arms: Disitamab Vedotin +RC148
Drug: RC148 — 20mg/kg, intravenous infusion, once every 2 weeks
  Arms: Disitamab Vedotin +RC148
Drug: Albumin-bound Paclitaxone — 125 mg/m2,intravenous infusion, D1-8, every 3 weeks
  Arms: Albumin-bound Paclitaxone OR Albumin-bound Paclitaxone +Toripalimab
Drug: Toripalimab — 240mg,intravenous infusion, once every 3 weeks
  Other Names: JS001
  Arms: Albumin-bound Paclitaxone OR Albumin-bound Paclitaxone +Toripalimab

SUMMARY:
Evaluating the Efficacy of Disitamab Vedotin in Combination with RC148 Compared to Albumin-bound Paclitaxone Monotherapy or in Combination with Toripalimab for Subjects with HR-negative, HER2-low Expressing Unresectable Locally Advanced or Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study and sign the informed consent form
* Stage III unresectable locally advanced or Stage IV metastatic breast cancer.
* Subjects must be willing and able to provide a tumor tissue block and/or unstained pathology slides, with priority given to the most recent metastatic lesions that have not previously been subjected to radiotherapy. If this is not feasible or available, then a tumor tissue block (or fresh tissue sections) obtained from locally recurrent lesions should be provided. Freshly obtained tissue is preferred over archived tissue. The provided tissue will be used for biomarker testing and must be suitable for analysis of HER2 expression and PD-L1 expression
* Invasive breast tumor tissue has been confirmed as HER2 low expression by the central laboratory
* Invasive tumor tissue is negative for hormone receptors (HR), defined as immunohistochemistry (IHC) testing showing that the proportion of cells with positive nuclear staining for both ER and PgR in invasive cancer is less than 1%. For patients with weakly positive ER/PgR (1% to 10% of tumor cell nuclei positive), those who are not suitable for endocrine therapy after thorough evaluation by the investigator, and with approval from the sponsor after communication, may be included in this study
* For HR-negative, HER2-low expressing unresectable locally advanced or metastatic breast cancer: locally recurrent and unresectable or previously untreated metastatic breast cancer; or those who have completed curative treatment (excluding radiotherapy) (e.g., the date of surgery for the primary breast tumor or the last date of adjuvant therapy administration, whichever is later), with an interval of ≥6 months from the first documented local or distant disease recurrence. For subjects who received taxane drugs during the (neo)adjuvant therapy phase, there must be an interval of ≥12 months from the last taxane administration
* ECOG performance status of 0 or 1
* According to the RECIST v1.1 criteria, there must be at least one measurable lesion (for lesions that have previously been irradiated, if the lesion can be measured according to the RECIST v1.1 criteria and there is evidence of significant progression after radiotherapy, the lesion can be considered a target lesion)
* Expected survival of at least 12 weeks
* Hematologic and organ function criteria to be met within 7 days prior to the first dose of study medication (with normal values based on the clinical trial center's standards, and no blood transfusions, hematopoietic growth factors, albumin, or blood products within 14 days prior to the test):

Hemoglobin ≥ 90 g/L Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L Platelet count ≥ 100 × 10^9/L Total bilirubin ≤ 1.5 × upper limit of normal (ULN) or direct bilirubin ≤ ULN (for subjects with total bilirubin > 1.5 × ULN). Total bilirubin ≤ 3 × ULN (for subjects with Gilbert's disease) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN (if liver metastases are present) International normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN Creatinine clearance (CrCl) calculated by the Cockcroft-Gault formula ≥ 40 mL/min, or serum creatinine ≤ 1.5 × ULN Urine routine test shows urine protein < 2+; if urine protein ≥ 2+, the 24-hour urine protein quantification result must be < 1 g.

* Female subjects of childbearing potential who meet the following conditions:

A serum pregnancy test (with a minimum sensitivity of 25 mIU/mL or equivalent units of β-human chorionic gonadotropin [β-hCG]) must be negative within 7 days prior to the first dose of study intervention. Subjects with a false-positive result that is confirmed not to be pregnant are eligible to participate in the study.

Must agree to use contraception during the study and for at least 6 months after the last dose of study medication. No breastfeeding or egg donation within 6 months.

If sexual activity could lead to pregnancy, they must use at least one acceptable form of contraception from the time of informed consent until at least 6 months after the last dose of study medication.

* Male subjects of childbearing potential who meet the following conditions:

Must agree to abstain from donating sperm from the start of the study until at least 6 months after the last dose of study medication.

If having sexual intercourse with a person of childbearing potential that could lead to pregnancy, must consistently use at least one acceptable form of contraception throughout the study and for at least 6 months after the last dose of study medication.

If having sexual intercourse with a pregnant or breastfeeding partner, must use condoms from the time of informed consent until at least 6 months after the last dose of study medication.

* Capable of understanding the trial requirements and willing and able to comply with the trial and follow-up procedures.

Exclusion Criteria:

* Having previously received anti-HER2 treatment, including ADC (Antibody-Drug Conjugates).
* Having previously received immunotherapy, including anti PD-(L)1 or anti PD-(L)2 drugs, or drugs that directly target another stimulatory or co-inhibitory T-cell receptor (such as CD137, CTLA-4, OX-40) during the locally advanced or metastatic stage (except if the last administration was ≥12 months prior to recurrence or progression, using [neo]adjuvant anti PD-(L)1).
* Excluding subjects with brain metastases or leptomeningeal metastases. Subjects with treated brain metastases (surgery and/or radiotherapy) are eligible for inclusion if they meet the following criteria:

Subjects who have received treatment for brain metastases may be considered for participation in this study if they have not experienced disease progression as determined by imaging studies within 4 weeks prior to the first dose of study treatment.

They must have discontinued the use of corticosteroids or anticonvulsant therapy at least 14 days before the first dose of study

* Use of investigational drugs or undergoing major surgery within 4 weeks prior to the first dose of study medication
* Received or plan to receive live vaccines or attenuated live vaccines within 4 weeks prior to the first dose of study medication or during the study period
* History of allogeneic hematopoietic stem cell transplantation or organ transplantation
* Uncontrolled or significant cardiovascular or cerebrovascular disease, including (but not limited to):

Within 6 months prior to the first dose of study medication, any of the following occurred: congestive heart failure (NYHA Class III or IV), myocardial infarction, or cerebral infarction (except for lacunar infarction), pulmonary embolism, unstable angina, or the presence of arrhythmias requiring treatment at screening; Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, unclassified cardiomyopathy); A history of clinically significant QTc interval prolongation, second-degree type II atrioventricular block or third-degree atrioventricular block, or QTc interval (Fridericia's formula) > 470 msec (females) or > 450 msec (males); Atrial fibrillation (EHRA classification ≥ class 2b); Uncontrolled hypertension, as judged by the investigator to be unsuitable for participation in the study

* Presence of clinically uncontrollable third space fluid accumulation, such as large amounts of pleural effusion, pericardial effusion, or ascites that are associated with clinical symptoms or require symptomatic treatment.
* History of interstitial lung disease that requires treatment or current severe pulmonary disease, including but not limited to active pulmonary tuberculosis, interstitial lung disease, etc.
* A clear history of neurological or psychiatric disorders, either past or present, including epilepsy or dementia, etc.
* Toxicities from previous anti-cancer treatments have not yet recovered to grade 0-1 of the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0), except for alopecia, hyperpigmentation, or other conditions that the investigator deems do not increase the risk to the subject from treatment.
* Persistent grade ≥2 sensory or motor neuropathy.
* Active infections that require systemic treatment:

Active infections requiring systemic treatment within 7 days prior to the first dose, routine antimicrobial prophylaxis is allowed; Positive HIV test results; Patients with active hepatitis B or C (HBsAg positive with detectable HBV DNA levels above the upper limit of normal; HCVAb positive with detectable HCV RNA levels above the upper limit of normal).

* Having active autoimmune diseases within the past 2 years that require systemic treatment (such as corticosteroids or immunosuppressive drugs), except for replacement therapies (such as thyroid hormone, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency).
* Having other malignant tumors within 5 years prior to signing the informed consent form (except for effectively treated non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, stage I endometrial cancer, or other tumors that are considered cured).
* Known hypersensitivity or delayed-type allergic reactions to certain components of Disitamab Vedotin, Toripalimab, RC148, or albumin-bound paclitaxone, or similar drugs.
* According to the investigator's judgment, there are serious concomitant diseases that could endanger the subject's safety or affect the subject's ability to complete the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1

SECONDARY OUTCOMES:
PFS | From the first dose to the first documentation of disease progression or death, up to two years
  Progression-free survival is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first
DCR | 24 months
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1
OS | up to 5 years
  OS is the time from randomization to death due to any cause safety

CONTACTS AND LOCATIONS:
Locations (1):
- Cance Hosoltal Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China